CLINICAL TRIAL: NCT02230995
Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Metformin Extended Release (25 mg/1000 mg) Compared With the Free Combination of Empagliflozin and Metformin Extended Release Tablets in Healthy Subjects Following a High-fat, High-caloric Meal (an Open-label, Randomised, Single Dose, Crossover Trial)
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Metformin Extended Release Compared With Mono Compound Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.15; 2014-002016-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; empagliflozin

ARMS (2):
- Fixed dose combination (Experimental): Single dose empagliflozin/metformin
  Interventions: Drug: empagliflozin/metformin
- Single tablets combination (Active Comparator): single doses empagliflozin and metformin
  Interventions: Drug: metformin; Drug: empagliflozin

INTERVENTIONS:
Drug: metformin — single dose of metformin given as tablets
  Arms: Single tablets combination
Drug: empagliflozin/metformin — Single dose empagliflozin/metformin given as fixed-dose combination tablet
  Arms: Fixed dose combination
Drug: empagliflozin — single dose of empagliflozin given as tablet
  Arms: Single tablets combination

SUMMARY:
The purpose of this trial is to demonstrate bioequivalence of a newly developed fixed dose combination (FDC) tablet containing empagliflozin and metformin extended release compared to the free combination of empagliflozin and metformin extended release under fed conditions.

ELIGIBILITY:
Inclusion criteria:

- Healthy male and female subjects

Exclusion criteria:

- Any relevant deviation from healthy condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Biberach an der Riss, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, randomised, 2-way crossover trial with 2 treatments (T and R) and 2 treatment sequences (T_R and R_T). Trial drug administrations of the 2 single dose treatments were separated by a washout period of at least 7 days.
Groups:
- Fed 25mg+1000mg FDC/Single: Subjects received in period 1 a single dose of 25 mg empagliflozin/1000 mg metformin HCl XR (1 FDC tablet) with 240 mL of water after intake of a high-fat, high-caloric meal, followed in period 2 with a single dose of 25 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal.
  2 treatments separated by a wash-out period of at least 7 days.
- Fed 25mg+1000mg Single/FDC: Subjects received in period 1 a single dose of 25 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal, followed in period 2 with a single dose of 25 mg empagliflozin/1000 mg metformin HCl XR (1 FDC tablet) with 240 mL of water after intake of a high-fat, high-caloric meal.
  2 treatments separated by a wash-out period of at least 7 days.
Period: Period 1 + Washout
Arm/Group | Fed 25mg+1000mg FDC/Single | Fed 25mg+1000mg Single/FDC
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2 + Washout
Arm/Group | Fed 25mg+1000mg FDC/Single | Fed 25mg+1000mg Single/FDC
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fed 25mg+1000mg FDC/Single | Fed 25mg+1000mg Single/FDC | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.60 (9.30) | 32.00 (9.80) | 34.30 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz of Empagliflozin in Plasma
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 to the time of the last quantifiable concentration (AUC0-tz)
Time Frame: -1:00 hour(h) before the drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 4:00h, 5:00h, 6:00h, 7:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h and 72:00h after drug administration
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Groups:
- Fed 25mg+1000mg FDC: Subjects received a single dose of 25 mg empagliflozin/1000 mg metformin Hydrochloride (HCl) Extended release (XR) (1 Fixed dose combination (FDC) tablet) with 240 mL of water after intake of a high-fat, high-caloric meal.
- Fed 25mg+1000mg Single: Subject received a single dose of 25 mg empagliflozin (1 tablet) together with 1000 mg metformin HCl XR (2 tablets) with 240 mL of water after intake of a high-fat, high-caloric meal.
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
nmol·h/L | 5370 (14.9) | 5470 (16.0)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based on 2-sided 90% confidence intervals (CIs) for the ratios (test to reference treatment) of the adjusted geometric means (gMeans) of the primary endpoints, using an acceptance range of 80.00 to 125.00%; p < 0.00001, ANOVA; ANOVA model on the logarithmic scale including random effects for 'subjects within sequences' & fixed effect for 'sequence', 'period' & 'treatment'; Adjusted gMean ratio = 98.22, 90% CI 2-sided [96.11 to 100.39], Standard Deviation 5.0 — Relative bioavailability of empagliflozin was estimated by the ratios of the adjusted gMean of Fed 25mg+1000mg FDC divided by Fed 25mg+1000mg Single. Standard deviation is actually Intra individual geometric coefficient variation (gCV)

2. Primary Outcome: AUC0-tz of Metformin in Plasma
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable concentration
Time Frame: as for outcome 1
Population: Pharmacokinetic Set (PKS): This analysis set included all treated subjects that provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of the pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
ng·h/mL | 11000 (21.5) | 10800 (22.8)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.00001, ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean ratio = 102.14, 90% CI 2-sided [98.65 to 105.76], Standard Deviation 7.9 — Relative bioavailability of metformin was estimated by the ratios of the adjusted gMean of Fed 25mg+1000mg FDC divided by Fed 25mg+1000mg Single. Standard deviation is actually Intra individual geometric coefficient variation (gCV)

3. Primary Outcome: Cmax of Empagliflozin in Plasma
Description: Maximum measured concentration of empagliflozin in plasma (Cmax)
Time Frame: as for outcome 1
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
nmol/L | 590 (19.9) | 597 (19.5)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.00001, ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean ratio = 98.70, 90% CI 2-sided [93.51 to 104.17], Standard Deviation 12.3 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Cmax of Metformin in Plasma
Description: Maximum measured concentration of the metformin in plasma
Time Frame: as for outcome 1
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
ng/mL | 1120 (23.0) | 1060 (24.9)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.00001, ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean ratio = 105.69, 90% CI 2-sided [100.78 to 110.84], Standard Deviation 10.9 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: AUC0-infinity of Empagliflozin in Plasma
Description: Area under the concentration-time curve of empagliflozin in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity)
Time Frame: as for outcome 1
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol·h/L
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
nmol·h/L | 5460 (15.1) | 5550 (16.2)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean ratio = 98.32, 90% CI 2-sided [96.16 to 100.53], Standard Deviation 5.1 — Relative bioavailability of empagliflozin was estimated by ratios of adjusted geometric means (gMean) of Fed 25mg+1000mg FDC divided by Fed 25mg+1000mg Single. Standard deviation is actually Intra individual geometric coefficient variation (gCV)

6. Secondary Outcome: AUC0-infinity of Metformin in Plasma
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 1
Population: PKS set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Number analyzed (Participants) | 30 | 30
ng*h/mL | 11500 (20.2) | 11000 (22.7)
Statistical Analysis 1: Comparison: Fed 25mg+1000mg FDC vs Fed 25mg+1000mg Single; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gMean ratio = 104.66, 90% CI 2-sided [101.36 to 108.07], Standard Deviation 7.3 — Relative bioavailability of metformin was estimated by the ratios of the adjusted geometric means (gMean) of Fed 25mg+1000mg FDC divided by Fed 25mg+1000mg Single. Standard deviation is actually Intra individual geometric coefficient variation (gCV)

ADVERSE EVENTS:
Time Frame: From first drug administration up to 13 days after last drug administration, ie., upto 20 days.
Arm/Group | Fed 25mg+1000mg FDC | Fed 25mg+1000mg Single
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fed 25mg+1000mg FDC (N=30) | Fed 25mg+1000mg Single (N=30)
Nasopharyngitis (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes